CLINICAL TRIAL: NCT05387070
Title: PaTHway CHINA TRIAL: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Trial, With an Open-Label Extension, Investigating the Safety, Tolerability and Efficacy of TransCon PTH Administered Subcutaneously Daily in Adults With Hypoparathyroidism
Brief Title: PaTHway CHINA TRIAL: A Trial to Investigating the Safety, Tolerability and Efficacy of TransCon PTH in Adults With Hypoparathyroidism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Visen Pharmaceuticals (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCP-306; CTR20212047 (Other: Center for drug evaluation, NMPA)
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hypoparathyroidism; Parathyroid Hormone Deficiency; Endocrine System Diseases; Parathyroid Diseases
Keywords: Hypoparathyroidism; TransCon PTH; Parathyroid Hormone deficiency; PTH1-34
MeSH Terms: conditions — Hypoparathyroidism; Endocrine System Diseases; Parathyroid Diseases

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 3:1 to receive either TransCon PTH or placebo:
  * TransCon PTH 18 μg/day* , co-administered with SoC
  * Placebo for TransCon PTH (excipient solution) 18 μg/day, co-administered with SoC
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TransCon PTH (Experimental): TransCon PTH at a starting dose of 18 mcg delivered once daily by subcutaneous injection
  Interventions: Drug: TransCon PTH
- placebo (Placebo Comparator): Placebo for TransCon PTH at a starting dose of 18 mcg delivered once daily by subcutaneous injection
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: TransCon PTH — TransCon PTH is supplied as a solution with a concentration of 0.3 mg PTH(1-34)/mL in a single-patient-use prefilled pen intended for SC injection.
  Arms: TransCon PTH
Drug: placebo — Placebo is supplied as a solution containing the formulation buffer for TransCon PTH in a single-patient-use prefilled pen intended for subcutaneous injection.
  Arms: placebo

SUMMARY:
This study is limited to conduct in China only. The primary objective is to assess the treatment effect of daily TransCon PTH on serum calcium (sCa) levels within the normal range and stopping from therapeutic doses of active vitamin D (calcitriol) or active vitamin D analogue (alfacalcidol) and calcium at 26 weeks of treatment. All subjects will start with 18 mcg of study drug and will be individually and progressively titrated to an optimal dose over a 26-week double blind period, followed by an open label extension period up to 156 weeks. TransCon PTH or placebo will be administered as a subcutaneous injection using a pre-filled injection pen. Neither trial participants nor their doctors will know who has been assigned to each group. After the 26 weeks, participants will continue in the trial as part of a long-term extension study. During the extension, all participants will receive TransCon PTH, with the dose adjusted to their individual needs.

DETAILED DESCRIPTION:
Not Provided

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, ≥18 years of age
2. Subjects with postsurgical chronic HP, or auto-immune, genetic, or idiopathic HP for at least 26 weeks. Diagnosis of HP is established based on historic hypocalcemia in the setting of inappropriately low (below the ULN of local laboratory) serum PTH levels.
3. Requirement for doses of SoC (e.g., calcitriol, alfacalcidol, calcium supplements) at or above a minimum threshold:

   • requirement for a dose of calcitriol ≥0.5 μg/day, or alfacalcidol ≥1.0 μg/day and (elemental) calcium ≥800 mg/day (e.g., calcium citrate, calcium carbonate etc.) for at least 12 weeks prior to Screening. In addition, the dose of calcitriol, or alfacalcidol, and calcium should be stable for at least 5 weeks prior to Screening
4. Optimization of supplements prior to randomization to achieve the target serum levels of:

   * 25(OH) vitamin D levels of 10-100 ng/mL (25-250 nmol/L) and
   * Magnesium level in the normal range, or just below the normal range i.e.: ≥1.3 mg/dL (0.53 mmol/L) and
   * Albumin-adjusted sCa level in the normal range, or just below the normal range, i.e.: 7.8-10.6 mg/dL (or 1.95-2.64 mmol/L)
5. The subject demonstrates a 24-hour uCa excretion of ≥125 mg/24h (on a sample collected within 52 weeks prior to Screening or during the Screening Period)
6. BMI 17- 40 kg/m2 at Screening
7. If ≤25 years of age, radiological evidence of epiphyseal closure based on X-ray of non-dominant wrist and hand
8. Thyroid-stimulating hormone (TSH) within normal laboratory limits within the 6 weeks prior to Visit 1; if on suppressive therapy for a history of thyroid cancer, TSH level must be ≥0.2 mIU/L
9. If treated with thyroid hormone replacement therapy, the dose must have been stable for at least 5 weeks prior to Screening
10. eGFR ≥30 mL/min/1.73 m2 during Screening
11. Able to perform daily SC self-injections of study drug (or have a designee to perform injections) via a pre-filled injection pen
12. Able and willing to provide written and signed ICF in accordance with GCP

Exclusion Criteria:

1. Impaired responsiveness to PTH (pseudohypoparathyroidism) which is characterized as PTH-resistance, with elevated PTH levels in the setting of hypocalcemia
2. Any disease that might affect calcium metabolism or calcium-phosphate homeostasis or PTH levels other than HP, such as active hyperthyroidism; Paget disease of bone; severe hypomagnesemia; type 1 diabetes mellitus or poorly controlled type 2 diabetes mellitus (HbA1C >9%, documented HbA1C result drawn within 12 weeks prior to Screening is acceptable); severe and chronic liver, or renal disease; Cushing syndrome; multiple myeloma; active pancreatitis; malnutrition; rickets; recent prolonged immobility; active malignancy (other than low-risk well differentiated thyroid cancer or non-melanoma skin cancer); active hyperparathyroidism; parathyroid carcinoma within 5 years prior to Screening; acromegaly;or multiple endocrine neoplasia
3. High risk thyroid cancer within 2 years, requiring suppression of TSH <0.2 mIU/L
4. Long term use of loop diuretics, phosphate binders (other than calcium supplements), digoxin, lithium, methotrexate, biotin >30 µg/day, or systemic corticosteroids (other than as replacement therapy)
5. Use of thiazide diuretic within 4 weeks prior to the 24-hour urine collection scheduled to occur within 1 week prior to Visit 1
6. Use of PTH-like drugs (whether commercially available or through participation in an investigational trial), including PTH (1-84), PTH (1-34), or other N-terminal fragments or analogs of PTH or PTH-related protein, within 4 weeks prior to Screening
7. Use of other drugs known to influence calcium and bone metabolism, such as calcitonin, fluoride tablets (>0.5 mg/day), strontium, or cinacalcet hydrochloride, within 12 weeks prior to Screening
8. Use of osteoporosis therapies known to influence calcium and bone metabolism, i.e., bisphosphonate (oral or intravenous [IV]), denosumab, raloxifene, or romosozumab therapies within 2 years prior to Screening
9. Non-hypocalcemic seizure disorder with a history of a seizure within 26 weeks prior to Screening
10. Increased risk for osteosarcoma, such as those with Paget's disease of bone or unexplained elevations of alkaline phosphatase, hereditary disorders predisposing to osteosarcoma, or with a prior history of substantial external beam or implant radiation therapy involving the skeleton
11. Pregnant or lactating women
12. Male who has a female partner who intends to become pregnant or is of childbearing potential and is unwilling to use adequate contraceptive methods during the trial
13. Diagnosed drug or alcohol dependence within 3 years prior to Screening
14. Disease processes that adversely affect gastrointestinal absorption, including but not limited to short bowel syndrome, significant small bowel resection, gastric bypass, tropical sprue, active celiac disease, active ulcerative colitis, active Crohn's disease, gastroparesis and AIRE gene mutations with malabsorption
15. Severe cardiac disease within 26 weeks prior to Screening including but not limited to congestive heart failure, myocardial infarction, severe or uncontrolled arrhythmias, bradycardia (resting heart rate <48 beats/minute, unless chronic and asymptomatic), symptomatic hypotension or systolic BP <80 mm Hg or diastolic <40 mm Hg or poorly controlled hypertension (systolic BP >165 mm Hg or diastolic >95 mm Hg). In the absence of a prior history of hypertension, an isolated BP >165/95 mm Hg in the setting of white coat hypertension/anxiety may not be exclusionary and a measurement can be repeated prior to randomization
16. Cerebrovascular accident within 5 years prior to Screening
17. Within 26 weeks prior to Screening: acute colic due to nephrolithiasis, or acute gout. Subjects with asymptomatic renal stones are permitted
18. Participation in any other interventional trial in which receipt of investigational drug or device occurred within 8 weeks (or within 5.5 times the half-life of the investigational drug) (whichever comes first) prior to Screening
19. Any disease or condition that, in the opinion of the investigator, may require treatment or make the subject unlikely to fully complete the trial, or any condition that presents undue risk from the investigational product or procedures, including treated malignancies that are likely to recur within the approximate 3.5-year duration of the trial
20. Known allergy or sensitivity to PTH or any of the excipients [metacresol, mannitol, succinic acid, NaOH/(HCl)]
21. Likely to be non-compliant with respect to trial conduct
22. Any other reason that in the opinion of the investigator would prevent the subject from completing participation or following the trial schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2026-01-08 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects who meet primary efficacy endpoint at 26 weeks of treatment | 26 weeks
  The proportion of subjects with albumin-adjusted sCa within the normal range, and independence from active vitamin D, and independence from therapeutic doses of calcium (i.e., taking calcium supplements ≤600 mg/day), and no increase in prescribed study drug within 4 weeks prior to Week 26 visit

SECONDARY OUTCOMES:
Change from baseline in HPES Symptom - Physical Domain score | 26 weeks
  Change from baseline in Hypoparathyroidism Patient Experience Scale (HPES) Symptom - Physical Domain score, a disease-specific patient reported outcome, at 26 weeks of treatment

OTHER OUTCOMES:
Change from baseline in HPES Symptom - Cognitive Domain score | 26 weeks
  Change from baseline in Hypoparathyroidism Patient Experience Scale (HPES) Symptom - Cognitive Domain score, a disease-specific patient reported outcome, at 26 weeks of treatment
Change from baseline in HPES Impact - Physical Functioning Domain score | 26 weeks
  Change from baseline in Hypoparathyroidism Patient Experience Scale (HPES) Impact - Physical Functioning Domain score, a disease-specific patient reported outcome, at 26 weeks of treatment
Change from baseline in HPES Impact - Daily Life Domain score | 26 weeks
  Change from baseline in Hypoparathyroidism Patient Experience Scale (HPES) Impact - Daily Life Domain score, a disease-specific patient reported outcome, at 26 weeks of treatment
Change from baseline in SF-36 Physical Functioning subscale score | 26 weeks
  Change from baseline in the 36-item Short Form Survey (SF-36) Physical Functioning subscale score, a generic health survey, at 26 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Weibo Xia, MD, Principal Investigator — Department of endocrinology, Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No